CLINICAL TRIAL: NCT03415373
Title: Clinical Evaluation of Healthy Subjects Receiving Intradermal Saline Using the Microneedle Adapter (Model UAR-2S)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microdermics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UAR-CLIN-001
Record Dates: First submitted 2018-01-18; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Intradermal Injection
MeSH Terms: interventions — Needles; Syringes

STUDY DESIGN:
Intervention Model Description: Subjects will be first randomized to receive each of the injection (A, B, C, and D) in each of the 3 visits of the study, according to the block randomization scheme produced by inVentiv. The following sequences will be used: 1st (upper right location), 2nd (lower right location), 3rd (upper left location) and 4th lower left location) where:
  A. Investigational device with 50 μL saline B. Control device with 50 μL saline C. Investigational device with 100 μL saline D. Control device with 100 μL saline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Each subject will undergo ID administration by Microneedle Adapter (Model UAR-2S) and hypodermic needle + syringe of 100 μL injectable saline into 3 different regions: the inner forearm, the deltoid and the thigh, at three (3) study visits. A total of 4 injections (2 x 50 μL saline and 2 x 100 μL saline) will be administered to each study participant in the injection sites (2 injections per inner forearm/deltoid/thigh and 2 injection per device).
  Interventions: Device: Microneedle Adapter (Model UAR-2S); Device: Hypodermic needle + syringe

INTERVENTIONS:
Device: Microneedle Adapter (Model UAR-2S) — Investigational device
Device: Hypodermic needle + syringe — Control device

SUMMARY:
Microdermics Inc. is a British Columbia-based Canadian incorporation primarily focusing on microneedle-based painless and effective drug delivery systems.The Microneedle Adapter (model UAR-2S) is a single-use disposable medical device intended to provide a mechanism for intradermal bolus fluid delivery when used with a standard syringe with a Luer-lock tip connection. The Microneedle Adapter consists of a single-use gold-coated metallic microneedle integrated within the microneedle adapter with fluidic connections to a standard Luer syringe mount. The primary function of the Microneedle Adapter is to guide the microneedle into the skin in a controlled manner for successful insertion passing the stratum corneum layer. The fluid loaded onto the syringe can then be injected precisely intradermally into the skin.The primary objective of this study is to evaluate the performance of the Microneedle Adapter in healthy subjects in 3 different injection sites. Pain perception of the Microneedle Adapter will be a key secondary outcome, compared with the control device.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 19-65 years old inclusive, non-smoker (no use of tobacco products within 3 months prior to screening)
2. Able to understand the informed consent form and willing to participate in study
3. Intact skin at the sites of injection
4. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive method throughout the study and for 30 days after the last study drug administration:

   1. intra-uterine contraceptive device placed at least 4 weeks prior to study drug administration;
   2. male condom with intravaginally applied spermicide starting at least 14 days prior to study drug administration;
   3. hormonal contraceptives starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study;
   4. sterile male partner (vasectomized since at least 6 months).

Exclusion Criteria:

1. Fear or anxiety of needles, or needle phobia
2. Known sensitivity to nickel
3. Presence of a skin condition at the treatment are that may affect the configuration or thickness of the dermal layer (e.g. plaque psoriasis)
4. Permanent makeup/tattoo/body piercing or other markings in the treatment area that would impact the ability to assess adverse events (e.g. erythema) following ID administration
5. Use of medication that may affect the mechanical properties of the skin in the treatment area (e.g. prolonged use of a steroids, analgesics or other non-steroidal inflammatory drugs)
6. Any implantable metal device in the treatment area
7. Any surgical procedure, or other invasive or non-invasive method of skin therapy hair removal or filers or Botox in the treatment area, performed in the past 1 months (in the treatment area).
8. Any form of suspicious lesion on the treatment area
9. Hypertrophic scarring, keloids, abnormal wound healing, as well as very dry and fragile skin.
10. Any infection/abscess/pain in treatment area
11. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash
12. History of skin allergy or hypersensitivity
13. History of easy bruising
14. Actively taking antibiotics for an infection
15. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
16. Any other condition that would exclude the subject study participation according to the Investigator's clinical judgment
17. Concurrent participation in any other clinical study
18. Unable to understand the informed consent
19. Unable to verbally communicate in English or French
20. If female, pregnant, suspected or planning to become pregnant or breast-feeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of the Microneedle Adapter in the inner forearm | 1 day
  Consistency of injected fluid volume by gravimetric technique
Evaluate the performance of the Microneedle Adapter in the deltoid | 1 day
  Consistency of injected fluid volume by gravimetric technique
Evaluate the performance of the Microneedle Adapter in the thigh | 1 day
  Consistency of injected fluid volume by gravimetric technique

SECONDARY OUTCOMES:
Evaluate pain perception of the Microneedle Adapter vs. the control device | 1 day (post needle injection and post fluid injection)
  Assessment of pain intensity using Numeric Rating Scale (NRS), a verbal 0-10 point scale where 0 means no pain and 10 means worst possible pain
Collection and evaluation of adverse events [safety and tolerability] | 2 weeks
  Events will be reported by severity and causality
Assessment of contact dermatitis using Draize Scale [safety and tolerability] | 2 weeks
  Draize scale has 4 components (Hemorrhage/petechiae, Erythema, Edema, Pruritus) with scores 0 up to 5, where 5 indicates worst event
Assess end-user satisfaction in using the Microneedle Adapter and obtain feedback on the device's design | 2 weeks
  Assessment of end-user usability using the modified System Usability Scale (mSUS), a 10-question scale producing a normalized score 0 to 100, where 0 indicates high user dissatisfaction and 100 indicates high user satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — inVentiv Health Clinique
Locations (1):
- inVentiv Health Clinique, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided